CLINICAL TRIAL: NCT02322723
Title: Real Life Evaluation of Rheumatoid Arthritis Patients in Israel Treated With HUMIRA
Acronym: ORIENT
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-987
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Adalimumab; real life; RA; Humira; Rheumatoid Arthritis; effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderately to severely active RA patients: Moderately to severely active RA patients aged 18 years or older, both male and female

SUMMARY:
In Israel, data is lacking regarding the long-term effectiveness of Adalimumab in outpatient real life setting. Moreover, the association between long-term effectiveness of Adalimumab and patients' functional status as well as cultural aspects of sick leaves and visits to physician's clinics has not been demonstrated in this population. This study will collect the required data in real life settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible to Adalimumab treatment according to the Israeli National Health Basket and for whom a decision of initiating Adalimumab has already been taken. Patients that are naïve to Adalimumab therapy, that have been prescribed adalimumab in accordance to physician's clinical decision and according to local guidelines, up to 30 days prior to screening.
2. Patient has performed tuberculosis (TB) screening and treatment according to national guidelines for TB screening prior to anti Tumor Necrosis Factor (anti-TNF) treatment.
3. Patient has been diagnosed with Rheumatoid Arthritis (RA) and has disease duration < 3 years.
4. Patient has moderately to severely active RA defined by Disease Activity Score (DAS) (moderately (3.2 ≤ DAS ≤ 5.1) severely (DAS ≥5.1))
5. Patient is able to sign written informed consent.
6. Patient is treated with Methotrexate (MTX) alone or in combination with other Disease Modifying Antirheumatic Drugs (DMARDs)
7. Patient might have been treated with another anti-TNF inhibitor agent if discontinued due to secondary loss of efficacy or side effects.

Exclusion Criteria:

1. Patient with known hypersensitivity to Adalimumab, or any of its components.
2. Patients suffering from serious infection, latent TB or other conditions prohibiting the use of Adalimumab.
3. Patient had previous non-response to an anti-TNF agent.
4. Patients currently treated with other biologic therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderately to severely active Rheumatoid Arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who reached clinical response at 6 months | At 6 months
  Proportion of patients who reached Disease Activity Score (DAS)-28 of less than 2.6 or a good DAS response compared to the score on Day 0.

SECONDARY OUTCOMES:
Proportion of patients who reached clinical response at 24 months | At 24 months
  Proportion of patients who reached Disease Activity Score (DAS)-28 of less than 2.6 or a good DAS response compared to the score on Day 0.
Change in patient's functional status | Up to 24 months
  Proportion of patients reaching HAQ <= 0.5
Change in frequency of sick leave episodes | Up to 24 months
  Change in frequency of sick leave episodes
Change in frequency of outpatient clinic visits | Up to 24 months
  Change in frequency of outpatient clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Dina Meyuhas, PhD, Study Chair — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com/